CLINICAL TRIAL: NCT00494715
Title: A Prospective, Randomized, Probe Trial to Evaluate Whether,at Comparable Blood Pressure Control,Combined Therapy With ACEI BEN and ARB VAL Reduces Progression to ESRD More Effectively Than BEN or VAL Alone in High Risk Patients With Type 2 Diabetes and Overt Nephropathy
Brief Title: Preventing ESRD in Overt Nephropathy of Type 2 Diabetes
Acronym: VALID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VALID; 2006-005951-14 (EudraCT Number)
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — benazepril; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Benazepril (Experimental)
  Interventions: Drug: Benazepril
- valsartan (Experimental)
  Interventions: Drug: Valsartan
- benazepril/valsartan (Experimental)
  Interventions: Drug: Benazepril/Valsartan

INTERVENTIONS:
Drug: Benazepril — Patients satisfying the inclusion/exclusion criteria will be randomly given equivalent doses (half the standard doses recommended by the manufacturer for blood pressure control) of benazepril (10 mg/day) or valsartan (160 mg/day) or one fourth of the standard doses of both agents in combination (benazepril 5 mg/day and valsartan 80 mg/day).If well tolerated, treatment will be up-titrated to full dose of benazepril (20 mg/day) or valsartan (320 mg/day) or one half of the standard doses of both agents in combination (benazepril 10 mg/day and valsartan 160 mg/day).
  Arms: Benazepril
Drug: Valsartan — Patients satisfying the inclusion/exclusion criteria will be randomly given equivalent doses (half the standard doses recommended by the manufacturer for blood pressure control) of benazepril (10 mg/day) or valsartan (160 mg/day) or one fourth of the standard doses of both agents in combination (benazepril 5 mg/day and valsartan 80 mg/day).If well tolerated, treatment will be up-titrated to full dose of benazepril (20 mg/day) or valsartan (320 mg/day) or one half of the standard doses of both agents in combination (benazepril 10 mg/day and valsartan 160 mg/day).
  Arms: valsartan
Drug: Benazepril/Valsartan — Patients satisfying the inclusion/exclusion criteria will be randomly given equivalent doses (half the standard doses recommended by the manufacturer for blood pressure control) of benazepril (10 mg/day) or valsartan (160 mg/day) or one fourth of the standard doses of both agents in combination (benazepril 5 mg/day and valsartan 80 mg/day).If well tolerated, treatment will be up-titrated to full dose of benazepril (20 mg/day) or valsartan (320 mg/day) or one half of the standard doses of both agents in combination (benazepril 10 mg/day and valsartan 160 mg/day).
  Arms: benazepril/valsartan

SUMMARY:
Nephropathy of type 2 diabetes is the leading cause of end stage renal disease (ESRD) world-wide and is associated with a dramatic excess cardiovascular morbidity and mortality. Two randomized trials found that angiotensin II receptor blockers (ARBs) reduce the incidence of ESRD by about 30%, but have no appreciable effects on cardiovascular mortality. Available data suggest that ACE inhibitors might be similarly renoprotective and even more cardioprotective, but large scale trials on ACE inhibitors, alone or combined with ARBs, in overt nephropathy of type 2 diabetes are missing.

This study will compare the effects, at comparable blood pressure control (systolic/diastolic <130/80 mmHg), of dual renin-angiotensin-system (RAS) blockade by half dose of benazepril and valsartan combination therapy as compared to single RAS blockade by benazepril or valsartan alone at full dose, 20 mg and 160 mg respectively, on ESRD and cardiovascular events in high-risk patients with type 2 diabetes and overt nephropathy, defined as serum creatinine >1.8 mg/dl and < 3.2 mg/dl and spot morning urine albumin to creatinine ratio >1000mg/g for the patients without previous ACE inhibitor and ARB therapy and >500mg/g for the patients with previous ACE inhibitor or ARB therapy and no specific contraindications to the study drugs. The relationships between renal and cardiovascular outcomes will also be evaluated.

102 patients will be treated for at least 3 years. At comparable blood pressure control, the study is expected to show a more effective reduction in ESRD and cardiovascular events with combined than with single drug ACE inhibitor or ARB therapy. As compared to ARB, ACE inhibitor therapy is expected to have a similar effect on ESRD, but a superior cardioprotective effect. Applied to clinical practice, the findings should help reducing renal and cardiovascular complications, and related treatment costs, of type 2 diabetes.

DETAILED DESCRIPTION:
Introduction Nephropathy of type 2 diabetes is the leading cause of end stage renal disease (ESRD). Currently, more than 50% of patients on renal replacement therapy in the US are diabetics. The yearly incidence of diabetics progressing to ESRD and the proportion of ESRD patients with diabetes is progressively increasing due to the progressively increasing prevalence of type 2 diabetes worldwide.

Two large, multinational trials in overt nephropathy of type 2 diabetes found that interruption of the renin angiotensin system (RAS) with angiotensin II receptor blockers (ARBs) reduces the incidence of ESRD by about 30%, but has no appreciable effects on cardiovascular mortality. On the basis of these findings, ARB therapy has become standard treatment of patients with type 2 diabetes and nephropathy. However, despite ARB treatment, about 7% of patients continue to progress to ESRD and 7% continue to die every year.

Large-scale randomized trials evaluating the nephro- and cardio-protective effects of RAS inhibition with angiotensin-converting enzyme (ACE) inhibitors in overt nephropathy of type 2 diabetes are missing. However, studies in patients with type 1 diabetic nephropathy showed that ACE inhibitor therapy may decrease progression to ESRD by 40% and cardiovascular mortality by about 50%. Similar studies in non diabetic chronic nephropathies. consistently found a 40-50% reduction in the risk of progression to ESRD with ACE inhibitors as compared to non-RAS inhibitor therapy. Moreover, a meta-analysis of studies including type 2 diabetic patients with different degree of renal involvement showed that ACE inhibitors and ARBs sheared a similar renoprotective effect, but only ACE inhibitors significantly decreased the cardiovascular mortality.

A recent trial in non diabetic nephropathies found that combined RAS inhibition with ARBs and ACE inhibitors decreases progression to ESRD by 50% as compared to ARB or ACE inhibition alone. Evidence that combined therapy more effectively than ACE inhibitor or ARB therapy alone reduces albuminuria or proteinuria in patients with type 2 diabetes, suggests that a similar renoprotective effect could be achieved also in overt nephropathy of type 2 diabetes. Indeed, short-term proteinuria reduction is a strong predictor of slower progression of renal disease and reduced cardiovascular mortality in the long term.

A randomized trial powered to detect a reduced incidence of ESRD or cardiovascular mortality with combined ARB and ACE inhibition as compared to ACE inhibition or ARB alone would require several thousands of patients. However, identifying high risk patients who may benefit the most of nephro- and cardio-protective therapy would allow to design an adequately powered trial with remarkably less patients. By using a Bayesian decision-tree analysis we identified, among patients included in the RENAAL study, a subgroup of high risk patients with a baseline serum creatinine of 1.8 mg/dl or more and spot morning urine albumin to creatinine ratio >1000mg/g or more. Of note, over 3.5 year follow-up, 70% of these high-risk patients progressed to ESRD despite ARB therapy. Thus, the incidence of ESRD was three-fold higher in high-risk patients (20%) than in the whole study group (6.8%). High risk patients with these clinical characteristics are therefore the ideal target for randomized clinical trials aimed to evaluate the effect of novel nephro- and, possibly, cardio-protective treatments in overt nephropathy of type 2 diabetes.

Thus, whether dual more than single drug RAS blockade reduces the need for renal replacement therapy in high risk patients with type 2 diabetes and whether ACE inhibitors shear with ARBs a similar or even superior beneficial effect in this typology of patients is worth investigating. This could be of clinical relevance in these terms: 1. Effective prevention of ESRD in people with type 2 diabetes is expected to translate in a remarkable reduction in costs for renal replacement therapy by chronic dialysis or kidney transplantation; 2. A better definition of the cost/effectiveness profile of different study treatments may help optimizing the allocation of available resources in order to achieve more effective prevention at lower costs. 3. The definition of individual risk profiles may allows identifying subjects at increased risk that may benefit the most of intensified treatment, which should translate in a further optimization of the use of available resources at population level. Moreover, in addition to verify whether dual RAS blockade by combined ACE inhibitor and ARB treatment more effectively than single drug RAS blockade may prevent progression to ESRD, the present study will offer the opportunity to compare the renoprotective effects of equivalent doses of ACE inhibitors or ARBs.

Aims Primary To evaluate whether, at comparable blood pressure control, dual RAS blockade with combined therapy with halved doses of benazepril (10 mg/day) and valsartan (160 mg/day) reduces the incidence of ESRD more effectively than single drug RAS blockade by full doses of valsartan (320 mg/day) given alone in high-risk patients with type 2 diabetes and overt nephropathy.

Secondary

* To evaluate whether, at comparable blood pressure control, dual RAS blockade with combined therapy with halved doses of benazepril (10 mg/day) and valsartan (160 mg/day) reduces the incidence of ESRD more effectively than single drug RAS blockade by full doses of benazepril (20 mg/day) given alone in high-risk patients with type 2 diabetes and overt nephropathy.
* To evaluate whether, at comparable blood pressure control, the effects of benazepril and valsartan therapy are similar or whether, alternatively, one of the two treatments offers a superior protective effect against the progression to ESRD in the above study population.
* To evaluate the effects of the three study treatments on the incidence of fatal and non-fatal cardiovascular events, doubling of baseline serum creatinine, GFR decline and proteinuria,
* To assess the relationships, in the study group as a whole and within each treatment group, between renal outcome variables (ESRD, doubling serum creatinine, GFR decline, proteinuria) and fatal and non-fatal cardiovascular events, between achieved blood pressure or metabolic control and renal and/or cardiovascular outcome variables and between achieved proteinuria reduction or residual follow-up proteinuria and renal and/or cardiovascular outcome variables.

Design This will be a multicenter, Prospective, Randomized, Open label, Blinded End point (PROBE) trial of 3-year treatment with halved doses of benazepril (10 mg/day) and valsartan (160 mg/day) given in combination, or full doses of both benazepril (20 mg/day), or valsartan (320 mg/day) given alone in 102 consenting patients >40 year old, with type 2 diabetes (WHO criteria), serum creatinine >1.8 mg/dl and < 3.5 mg/dl, spot morning urine albumin to creatinine ratio >1000mg/g for the patients without previous ACE inhibitor and ARB therapy and >500mg/g for the patients with previous ACE inhibitor or ARB therapy and no specific contraindications to the study drugs. Primary efficacy variable will be ESRD and primary comparison will be between the benazepril plus valsartan and valsartan alone groups. The analysis will have an 80% power to detect (p=0.05, two-side test) a 50% difference in ESRD incidence.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >40 years old;
* High-risk subjects with type 2 diabetes (WHO criteria);
* Serum creatinine concentration of 1.8 mg/dl or more (but less than 3.5 mg/dl);
* Urinary albumin to creatinine ratio >1000mg/g for the patients without previous ACE inhibitor and ARB therapy and >500mg/g for the patients with previous ACE inhibitor or ARB therapy (in spot morning urine)
* Legal capacity;
* Written informed consent.

Exclusion Criteria:

* Specific contraindications or history of hypersensitivity to the study drugs or other;
* Serum potassium ≥ 6 mEq/L despite diuretic therapy, and optimized metabolic and acid/base control;
* Bilateral renal artery stenosis;
* Previous history of allergy or intolerance, or evidence of immunologically-mediated renal disease, systemic diseases, cancer;
* Drug or alcohol abuse;
* Any chronic clinical conditions that may affect completion of the trial or confound data interpretation;
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial;
* Evidence of an uncooperative attitude;
* Any evidence that patient will not be able to complete the trial follow-up;
* Dual RAS blockade with an ACE inhibitor and an ARB.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Progression to ESRD (i.e. need for renal replacement therapy by chronic dialysis or renal transplantation) | 4 times a year

SECONDARY OUTCOMES:
Doubling of serum creatinine (versus baseline), Rate of GFR decline, Incidence of fatal and non-fatal cardiovascular events (stroke, acute myocardial infarction, sudden death), Albumin to creatinine ratio and 24-hour urinary protein excretion. | 4 times a year

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (15):
- Italy (14):
  - Hospital "Azienda Ospedaliera Ospedali Riuniti di Bergamo" - Unit of Diabetology, Bergamo, Bergamo
  - Clinical Research Center for Rare Diseases "Aldo e Cele Daccò", Ranica, Bergamo
  - Hospital "Bolognini", Seriate, Bergamo
  - Hospital "S.Marta e S.Venera", Acireale, Catania
  - Hospital "Vittorio Emanuele-Ferrarotto-Santo Bambino", Catania, Catania
  - Hospital " Casa Sollievo della Sofferenza" - Unit of Nephrology, San Giovanni Rotondo, Foggia
  - University "Federico II", Napoli, Napoli
  - Hospital "G:Mazzini", Teramo, Teramo
  - IRCCS San Raffaele - Unit of General Medicine, Milan
  - Hospital "Azienda Ospedaliera di Parma" - Unit of Nephrology, Parma
  - Hospital "Azienda Ospedaliera di Treviglio e Caravaggio" - Ambulatory of Ponte San Pietro, Ponte San Pietro
  - Hospital "Azienda Ospedaliera di Treviglio e Caravaggio" Unit of Diabetology and Metabolic Diseases, Romano di Lombardia
  - University - AUSL 1 - Institute of Medical Pathology, Sassari
  - Hospital "Azienda Ospedaliera di Treviglio-Caravaggio"Unit of Diabetology and Metabolic Diseases, Treviglio
- Clinical Department of Endocrinology, Diabetes and Metabolic Diseases University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Cohen DL, Townsend RR. Is there added value to adding ARB to ACE inhibitors in the management of CKD? J Am Soc Nephrol. 2009 Aug;20(8):1666-8. doi: 10.1681/ASN.2008040381. Epub 2008 Sep 5. PMID 18776118